CLINICAL TRIAL: NCT05151952
Title: Proton Therapy Medical Registry
Status: Recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: Proton
Record Dates: First submitted 2021-11-11; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Cancer, Therapy-Related
Keywords: Proton therapy Additional relevant MeSH terms: Neoplasms, Secondary Primary Neoplasms, Cancer
MeSH Terms: conditions — Neoplasms, Second Primary; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients receiving proton radiation therapy: Cancer patients receiving proton radiation therapy, Registry of cancer patients who receive proton radiation therapy to crack disease and toxicity outcomes.
  Interventions: Radiation: Other: Registry

INTERVENTIONS:
Radiation: Other: Registry — Registry of cancer patients who receive proton radiation therapy.

SUMMARY:
Clínica Universidad de Navarra Proton Therapy Unit is establishing a registry to capture the full radiation dosimetry delivered to the patient, baseline clinical data, and disease, toxicity and quality of life outcomes. The objectives are parameters prescribed and to have all patients treated at the proton therapy unit to be included in the registry to enable future analysis of treatment outcomes to assist in understanding, which patients can benefit from the use of protons.

DETAILED DESCRIPTION:
Proton based radiation therapy has considerable dosimetric advantages over the standard photon based external beam radiation therapy, with an increased cost. Now, the clinical advantages, however, may not be identified in general, even with the improved dose distributions. In a large-scale evaluation, in time of personalized/ precision medicine, the impact of dosimetric benefit int clinical benefit meds registration studies.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated at the proton center

Exclusion Criteria:

* Any other than what is supplied in the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients with proton therapy
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2050-04-01 (Estimated)

PRIMARY OUTCOMES:
Outcome Mesure | 20 years
  Clinical outcomes will be obtains from electronic chart including: images, blood test, pathology and clinical reports

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Clinica Universidad de Navarra, Madrid